CLINICAL TRIAL: NCT03480542
Title: The CentrAl VenouS Catheter Access DocumEntation (CASCADE) Study
Brief Title: Central Venous Access Study
Acronym: CASCADE
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: PRO2016-0711
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-12

CONDITIONS: Central Line Catheters

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to document clinicians variation in practice in comparison to standard guidelines by the Medical Center's approved Evidence-based Practice (EBP) guidelines, policies, and procedures for Central Venous Catheter(CVC), Peripherally Inserted Central Catheter (PICC), and Hemodialysis (HD catheters by way of a structured retrospective review of the Electronic Medical Record (EMR) system.

DETAILED DESCRIPTION:
This will be a single site retrospective (non-experimental) study utilizing the electronic medical record, both descriptive and correlational methods.

There will be two outcomes:

1. The outcomes associated with the management of Central Venous Catheter(CVC), Peripherally Inserted Central Catheter (PICC), and Hemodialysis (HD) Catheter in adherence with hospital approved Evidence-based Practice guidelines for Central Venous Catheter(CVC), Peripherally Inserted Central Catheter (PICC), and Hemodialysis (HD) Catheter.
2. The mechanical/technical, thrombotic, and other adverse outcomes (Heparin induced coagulopathy) associated with central venous catheters due to variation in insertion and management practices of Central Venous Catheter(CVC), Peripherally Inserted Central Catheter (PICC), and Hemodialysis (HD) Catheter.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients in Medical Intensive Care Unit (MICU), Coronary Care Unit (CCU), Cardiac Surgical Intensive Care Unit (CSICU), Surgical Intensive Care Unit (SICU) with either CVCs, PICCs, or HD catheters.

Exclusion Criteria:

• Pediatric (including neonates), obstetric and gynecology, medical-surgical, and oncology patients.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three hundred patient electronic medical records will be reviewed from the Critical Care Units (Medical Intensive Care Unit, Coronary Care Unit, Cardiac Surgical Intensive Care Unit, Surgical Intensive Care Unit).
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Douglas, DNP, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
. If the results of the trial are published, participants' identities will remain confidential. Publication resulting from this research will not contain any information that could potentially identify participants either directly or indirectly.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of catheters was the focus of the study and because some patients had multiple catheters places, the number of patients does not coincide with the number of catheters.
Groups:
- Number of Hemodialysis Catheters: Number of patient medical records with incidence of hemodialysis catheters
- Number of Peripherally Inserted Central Venous Catheters: Number of patient medical records with incidence of peripherally inserted central venous catheters (PICC)
- Number of Central Venous Catheters: Number of patient medical records with incidence of central venous catheters (CVC)
Period: Overall Study
Arm/Group | Number of Hemodialysis Catheters | Number of Peripherally Inserted Central Venous Catheters | Number of Central Venous Catheters
Started | 12 | 53 | 152
Completed | 12 | 53 | 152
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For this retrospective data collection, 217 medical records were reviewed and met study eligibility criteria, this corresponds to 178 patients who received catheters during hospitalization (note, one patient may receive more than one catheter during hospitalization).
Groups:
- Number of Patients Who Received Hemodialysis Catheters: Number of patients who received hemodialysis catheters were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedure (note, patients received more than one catheter during hospitalization).
- Number of Patients Who Received Peripherally Inserted Peripherally Inserted Central Venous Catheters: Number of patients who received Peripherally Inserted Central Venous Catheters (PICC) were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedures(note, patients received more than one catheter during hospitalization).
- Number of Patients Who Received Central Venous Catheters: Number of patients who patients who received Central Venous Catheters (CVC) were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedures (note, patients received more than one catheter during hospitalization).
- Total: Total of all reporting groups
Arm/Group | Number of Patients Who Received Hemodialysis Catheters | Number of Patients Who Received Peripherally Inserted Peripherally Inserted Central Venous Catheters | Number of Patients Who Received Central Venous Catheters | Total
Number analyzed (Participants) | 12 | 39 | 127 | 178
Age, Continuous [Mean (Full Range); unit: years] | 62.6 [24 to 88] | 68 [22 to 99] | 65.6 [21 to 96] | 65.9 [21 to 99]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7 | 16 | 82 | 105
  Female | 5 | 23 | 45 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Clinical Guidelines for Catheter Interventions and Management
Description: Number of medical records with documented mechanical/technical, thrombotic, and other adverse outcomes associated with use of CVCs, PICCs, and Hemodialysis (HD) catheters.
Time Frame: 1 year
Population: Medical charts of eligible patients were reviewed and the number of patient medical charts with documentation are summarized. Note, a single patient may have received multiple catheters placed during their hospitalization.
Measure: Number; unit: # of catheter-related incidents
Units Other Than Participants: # of placed catheters
Groups:
- Patients Who Received Hemodialysis Catheters: Medical records of patients who received hemodialysis catheters were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedures.
- Patients Who Received Peripherally Inserted Central Venous Catheters (PICC): Medical records of patients who received peripherally inserted central venous catheters were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedures.
- Patients Who Received Central Venous Catheters (CVC): Medical records of patients who received central venous catheters were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedures.
Arm/Group | Patients Who Received Hemodialysis Catheters | Patients Who Received Peripherally Inserted Central Venous Catheters (PICC) | Patients Who Received Central Venous Catheters (CVC)
Number analyzed (Participants) | 12 | 39 | 127
Number analyzed (# of placed catheters) | 12 | 53 | 152
# of catheter-related incidents
  Number of documented Catheter Insertion Attempts | 12 | 0 | 0
  Number of documented Radiological Confirmation of Placement | 11 | 15 | 0
  Number of documented Fluoroscopy | 4 | 0 | 152
  Number of documented indications for catheter-use | 12 | 0 | 0
  Number of documented department/unit locations for Catheter Insertion | 8 | 14 | 152
  Number of documented Personnel conducting insertion | 12 | 0 | 0
  Number of documented dressing changes | 2 | 0 | 0
  Number of documented mask used at dressing change | 0 | 0 | 0
  Number of documented procedures accessed for central lines | 0 | 0 | 0
  Number of documented Scrub the hub procedures | 0 | 0 | 0
  Number of documented Alcohol impregnated caps used | 0 | 0 | 0
  Number of documented CUROS caps used | 1 | 0 | 0
  Number of documented flushes with normal saline | 11 | 0 | 0
  Number of documented flushes with heparin lock | 12 | 0 | 0
  Number of documented syringe sizes used for flushing | 3 | 0 | 0

2. Secondary Outcome: Number of Documented Catheter Complications
Description: Number of medical records with documented complications associated with the use of CVCs, PICCs, and Hemodialysis (HD) catheters
Time Frame: 1 year
Population: Medical charts of eligible patients with HD, PICC, and CVC catheters were reviewed for catheter complications
Measure: Number; unit: # of catheter-related incidents
Units Other Than Participants: Number of placed catheters
Groups:
- Records of Patients Who Received Hemodialysis Catheters: Medical records of patients who received hemodialysis catheters were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedures.
- Records of Patients Who Received Peripherally Inserted Central Venous Catheter (PICC): Medical records of patients who received Peripherally Inserted Central Venous Catheters (PICC) were reviewed for documentation of variation in practice in comparison to standard guidelines, policies and procedures.
- Records of Patients Who Received Central Venous Catheters (CVC): Medical records of patients who received Central Venous Catheters (CVC) were reviewed for documentation of variation in practice in comparison to standard guidelines, policies, and procedures.
Arm/Group | Records of Patients Who Received Hemodialysis Catheters | Records of Patients Who Received Peripherally Inserted Central Venous Catheter (PICC) | Records of Patients Who Received Central Venous Catheters (CVC)
Number analyzed (Participants) | 12 | 39 | 127
Number analyzed (Number of placed catheters) | 12 | 53 | 152
# of catheter-related incidents
  Number of Documented Mechanical complication | 0 | 0 | 0
  Number of Documented Mechanical complication type | 0 | 0 | 0
  Number of Documented Infections Complication | 0 | 0 | 0
  Number of Documented Infection complication type | 0 | 0 | 0
  Number of Documented Thrombotic complication | 0 | 0 | 0
  Number of Documented Thrombotic type | 0 | 0 | 0
  Number of Documented Catheter dwell | 0 | 0 | 0
  Number of documented date of Line insertion | 12 | 53 | 152
  Number of documented time of Line insertion | 11 | 53 | 152
  Number of documented date of Line removal | 12 | 53 | 152
  Number of documented time of Line removal | 12 | 53 | 152

ADVERSE EVENTS:
Time Frame: This study collected retrospective data from patient medical charts specific to catheter complications within primary and secondary outcomes and results. Consequently, no further adverse events were collected.
Description: This study collected retrospective data from patient medical charts specific to catheter complications within primary and secondary outcomes and results. Consequently, no further adverse events were collected.
Groups:
- Number of Hemodialysis Catheters: Number of patient medical records with an incidence of hemodialysis catheters
- Number of Peripherally Inserted Central Venous Catheters (PICC): Number of patient medical records with an incidence of peripherally inserted central venous catheters
- Number of Central Venous Catheters (CVC): Number of patient medical records with an incidence of central venous catheters
Arm/Group | Number of Hemodialysis Catheters | Number of Peripherally Inserted Central Venous Catheters (PICC) | Number of Central Venous Catheters (CVC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study is an observational retrospective study with no intervention. The number of catheters was the focus of the study and because some patients had multiple catheters places, the number of patients does not coincide with the number of catheters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT03480542/Prot_SAP_000.pdf